CLINICAL TRIAL: NCT05486481
Title: A Multicenter Phase 1/2 Study of Venetoclax/Daratumumab/Dexamethasone for Previously Treated Systemic Light-Chain Amyloidosis With Translocation (11;14)
Brief Title: Venetoclax, Daratumumab, and Dexamethasone for Systemic Light-Chain Amyloidosis With Translocation (11;14) (ALTITUDE)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Industry sponsor unable to continue support
Sponsor: Alfred Chung, MD (Other)
Collaborators: Janssen Pharmaceuticals (Industry); AbbVie (Industry)
Responsible Party: Sponsor-Investigator, Alfred Chung, MD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22253; NCI-2022-05530 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: AL Amyloidosis; Light Chain (AL) Amyloidosis; Systemic Light Chain Disease
Keywords: Translocation
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Amyloidosis | interventions — venetoclax; Dexamethasone; Calcium Dobesilate; daratumumab; In Situ Hybridization; In Situ Hybridization, Fluorescence; Biological Assay

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Phase I (venetoclax, dexamethasone, daratumumab) (Experimental): All participants receive 400 mg venetoclax once a day (QD) on days 1-28 of each cycle. Depending on the number of DLTs reported for this dose-level, participants may also receive dexamethasone on days 1, 8, 15, and 22 of each cycle with or without daratumumab on days 1, 8, 15, and 22 of cycles 1-2, days 1 and 15 of cycles 3-6, then on day 1 of cycles thereafter. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Venetoclax; Drug: Dexamethasone; Drug: Daratumumab; Device: Cyclin D1 gene (CCDN1) /immunoglobulin heavy chain (IGH) fluorescence in situ hybridization (FISH) assay
- Phase II (venetoclax, dexamethasone, daratumumab) (Experimental): Participants will receive the RP2D of venetoclax QD on days 1-28 of each cycle, dexamethasone on days 1, 8, 15, and 22 of each cycle, and daratumumab on days 1, 8, 15, and 22 of cycles 1-2, days 1 and 15 of cycles 3-6, then on day 1 of cycles thereafter. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: Venetoclax; Drug: Dexamethasone; Drug: Daratumumab; Device: Cyclin D1 gene (CCDN1) /immunoglobulin heavy chain (IGH) fluorescence in situ hybridization (FISH) assay

INTERVENTIONS:
Drug: Venetoclax — Given orally (PO)
  Other Names: Venclexta
Drug: Dexamethasone — Given PO
  Other Names: Ozurdex
Drug: Daratumumab — Given Subcutaneously (SC)
  Other Names: Darzalex; Daratumumab SC
Device: Cyclin D1 gene (CCDN1) /immunoglobulin heavy chain (IGH) fluorescence in situ hybridization (FISH) assay — Lab test

SUMMARY:
This phase I/II trial tests the safety, side effects, and best dose of venetoclax, daratumumab, and dexamethasone for the treatment of systemic light-chain amyloidosis in patients with a deoxyribonucleic acid (DNA) abnormality called a translocation involving chromosomes 11 and 14, or "t(11;14)". Venetoclax works by attaching to a protein called Bcl-2, in order to kill cancer cells. Daratumumab works by binding to a target on the surface of cancer cells called Cluster of differentiation 38 (CD38). When daratumumab binds to CD38, it enables the immune system to find the cancer cell and kill it. Dexamethasone is a type of drug called a corticosteroid. A corticosteroid is a drug made of artificial steroid hormones, that are used to treat symptoms such as inflammation (swelling and irritation to a part of the body). The combination of these medications may more effectively treat patients with systemic light-chain amyloidosis and t(11;14).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum-tolerated dose (MTD)/ the recommended phase 2 dose (RP2D) of venetoclax (VEN) with or without daratumumab subcutaneous (DARA SC) and dexamethasone (DEX), in previously treated light chain (AL) amyloidosis (PTAL) participants with t(11;14). (Phase I).

II. To evaluate the efficacy of the combination VEN/DARA SC and DEX as measured by Complete Hematologic Response (CHR rate) in PTAL participants with t(11;14). (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of VEN/DARA SC, and DEX in the treatment of PTAL participants with t(11;14). (Phase I) II. To evaluate the efficacy of VEN/DARA SC and DEX in the treatment of PTAL participants with t(11;14) as measured by overall hematologic response rate (ORR), progression free survival (PFS), overall survival (OS), organ response rate (orRR), major organ deterioration PFS (MOD-PFS), time to complete response (TTCR), duration of response (DOR), and time to new treatment (TTNT). To evaluate safety of VEN/DARA SC and DEX in the treatment of PTAL participants with t(11;14). (Phase II) IV. To evaluate the death rate, therapy-related death rate, infection rate, and cardiac event rate, in the VEN/DARA SC and DEX arm and the DARA SC and DEX arm. (Phase II).

EXPLORATORY OBJECTIVES:

I. To evaluate the feasibility of performing M protein detection by MALDI TOF mass spectrometry on the EXENT® system on serum and urine participant-samples collected by each site during the first 6 months of the study.

II. To evaluate the agreement between MALDI TOF mass spectrometry results by the EXENT® system and standard serologic and urine measures of disease after the enrollment for both phase 1 and 2 has been complete.

III. To evaluate the complete response (CR) rate, ORR, PFS, MOD-PFS, OS, OrRR, TTCR, TTNT and DOR separated by participants who are minimal residual disease (MRD) negative versus positive by EXENT®.

IV. To evaluate the CR rate, overall hematologic response rate (ORR), progression-free survival (PFS), major organ deterioration PFS (MOD-PFS), overall survival (OS), organ response rate (OrRR), time to complete response (TTCR), time to next treatment (TTNT) and duration of response (DOR) and relationship to light-chain glycosylation patterns over time by EXENT®.

OUTLINE: This is a phase I, dose-escalation study of venetoclax followed by a phase II study. If dose level 3 (VEN/DARA SC and DEX) is not the recommended phase 2 doses/maximum tolerated dose in phase 1, the study will not open to phase 2.

PHASE I: All participants receive venetoclax orally (PO) once daily (QD) on days 1-28 of each cycle. Depending on dose-level assignment, participants may also receive dexamethasone PO on days 1, 8, 15, and 22 of each cycle with or without daratumumab SC on days 1, 8, 15, and 22 of cycles 1-2, days 1 and 15 of cycles 3-6, then on day 1 of cycles thereafter. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

PHASE II: Participants receive venetoclax PO QD on days 1-28 of each cycle, dexamethasone PO on days 1, 8, 15, and 22 of each cycle, and daratumumab SC on days 1, 8, 15, and 22 of cycles 1-2, days 1 and 15 of cycles 3-6, then on day 1 of cycles thereafter. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 30 days and then every 3 months until the last participant on the study completes 2 years of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years
2. Histopathological diagnosis of amyloidosis based on detection by immunohistochemistry (IHC) and polarizing light microscopy of green bi-refringent material in Congo red-stained tissue specimens (in an organ other than bone marrow) or characteristic electron microscopy appearance.

   *Considerations for specific populations where other types of amyloidosis may be encountered:

   **For male subjects 70 years of age or older who have cardiac involvement only, and patients of African descent (black subjects), mass spectrometry typing of AL amyloid in a tissue biopsy is recommended to rule out other types of amyloidosis such as age-related amyloidosis or hereditary amyloidosis (ATTR mutation)
3. Presence of t(11;14) on bone marrow plasma cells (BMPC) by fluorescence in-situ hybridization (FISH), performed at the University of California San Francisco (UCSF) cytogenetics laboratory
4. >= 1 prior line of therapy for the treatment of systemic AL amyloidosis.

   *Note: Induction with only autologous stem cell transplant is considered 1 line of therapy. Steroid monotherapy treatment will not be counted as 1 prior line of therapy per National Comprehensive Cancer Network (NCCN) guidelines. Patients are not required to having progressed from the prior line of therapy
5. No prior CD38-directed antibody treatment OR If the patient previously received CD38-directed antibody treatment, the patient achieved >= partial response (PR) and did not progress while on CD38-directed antibody therapy. Progression on CD38-directed antibody treatment will be defined as progressive disease while on therapy or within 60 days of last dose.

   * Note: If the patient's last prior treatment included daratumumab and the patient relapsed (and does not meet the exclusion criteria as outlined in exclusion criterion #1) after cessation of treatment, a 3-month wash-out from CD38 antibody treatment is required. No washout period for DARA is deemed necessary when patients are already on DARA-based treatment and the treatment regimen needs to be stopped due to hematologic very good partial response (VGPR) or PR (suboptimal response) or non-DARA-related toxicity.
6. Measurable disease of light chain amyloidosis as defined by at least ONE of the following:

   1. Serum M-protein >= 0.5 g/dL by protein electrophoresis (routine serum protein electrophoresis and immunofixation (IFE) performed at a local laboratory),
   2. Serum free light chain >= 40mg/L with an abnormal kappa:lambda ratio or
   3. The difference between involved and uninvolved free light chains (dFLC) >= 20 mg/L.
7. One or more organs impacted by AL amyloidosis according to consensus guidelines.
8. Eastern Cooperative Oncology Group (ECOG) performance status =< 2.
9. Pretreatment clinical laboratory values meeting the following criteria during the Screening Phase (within 1 day of C1D1):

   1. Absolute neutrophil count >= 1.0 × 10^9/L without growth factor support for 7 days (14 days if pegfilgrastim).
   2. Hemoglobin level >= 8.0 g/dL (>= 5 mmol/L).
   3. Platelet count >= 100 × 10^9/L without transfusion for 14 days.
   4. Alanine aminotransferase level (ALT) =< 2.5 times the upper limit of normal (ULN).
   5. Aspartate aminotransferase (AST) =< 2.5 times the ULN.
   6. Total bilirubin level =< 3 × ULN except for subjects with Gilbert syndrome, in which case direct bilirubin =< 2 × ULN.
   7. Creatinine clearance of ≥ 30 mL/min based upon Cockcroft-Gault formula calculation or a 24-hour urine collection.
10. Patients must have completed other systemic therapy >= 14 days or investigational drug/vaccine >= 28 days prior to treatment, focal radiation therapy >= 14 days, surgery (other than biopsies) >= 21 days prior to treatment, and any autologous stem cell transplant (ASCT) >= 100 days prior to start of treatment.
11. Patients must not have received any medications or supplements which have been known to have some anti-amyloidogenic effect (such as: doxycycline; curcumin; prednisone; dexamethasone; epigallocatechin gallate) within 14 days prior to start of treatment.
12. Women of childbearing potential must commit to either abstain continuously from heterosexual sexual intercourse (if this is the preferred and usual lifestyle of the subject) or to use 2 methods of reliable birth control simultaneously. This includes one highly effective form of contraception (tubal ligation, intrauterine device, hormonal [birth control pills, injections, hormonal patches, vaginal rings or implants] or partner's vasectomy) and one additional effective contraceptive method (male latex or synthetic condom, diaphragm, or cervical cap). Contraception must begin 4 weeks prior to treatment and continue for 30 days after discontinuation of venetoclax or 3 months after discontinuation of DARA SC, whichever is longer. Reliable contraception is indicated even where there has been a history of infertility, unless due to hysterectomy or bilateral oophorectomy.
13. During the study and for 30 days after stopping VEN or 3 months after receiving the last dose of DARA SC, whichever is longer, a woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction.
14. A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control; e.g., either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository during and up to 30 days after discontinuation of VEN or 3 months after discontinuation DARA SC, whichever is longer. All men must also not donate sperm during the study and for 30 days after discontinuation of VEN or 3 months after discontinuation of DARA SC, whichever is longer.
15. Patients must have documentation of yearly flu vaccination and a pneumococcus vaccination. Note: If the patient is due for 2 doses of pneumococcus vaccination, patients must have documentation of having received one dose of vaccine. Live attenuated vaccines are not allowed
16. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Any prior hematologic progression to CD38 antibody therapy (regardless of presence of a response) while on treatment or within 90 days of the last dose. Hematologic progression is defined as any ONE of the following:

   1. From CR, any detectable monoclonal protein or abnormal free light chain ratio (the absolute concentration of the light chains must double)
   2. From PR, 50% increase in serum M protein to >0.5 g/dl or 50% increase in urine M protein to 4200 mg/day (a visible peak must be present)
   3. Free light chain increase of 50% to >100 mg/l
2. Prior exposure to BCL-2 inhibitors.
3. Intolerance to anti-CD38 antibody therapy, monoclonal antibodies, or hyaluronidase
4. Previous or current diagnosis of multiple myeloma by International Myeloma Working Group (IMWG) criteria, including the presence of lytic bone disease, plasmacytomas, >= 60% plasma cells in the bone marrow, or hypercalcemia.
5. Systemic AL amyloidosis from a lymphoma.
6. Any form of non-AL amyloidosis, including wild type or mutated (ATTR) amyloidosis.
7. Evidence of significant cardiovascular conditions as specified below:

   1. Troponin I >0.1 ng/ml and B-type natriuretic peptide (BNP) >700 pg/ml (cardiac stage 3B)
   2. Left ventricular ejection fraction (LVEF) <40%
   3. New York Heart Association (NYHA) classification IIIB or IV heart failure
   4. Heart failure that in the opinion of the investigator is on the basis of ischemic heart disease (e.g. prior myocardial infarction with documented history of cardiac enzyme elevation and electrocardiogram [ECG] changes) or uncorrected valvular disease and not primarily due to AL amyloid cardiomyopathy
   5. Inpatient admission to a hospital for unstable angina or myocardial infarction within the last 6 months prior to first dose or percutaneous cardiac intervention with recent stent within 6 months or coronary artery bypass grafting within 6 months
   6. For patients with congestive heart failure, cardiovascular-related hospitalizations within 4 weeks prior to Cycle 1 Day 1.
   7. Patients with a history of sustained ventricular tachycardia or aborted ventricular fibrillation or with a history of atrioventricular nodal or sinoatrial (SA) nodal dysfunction for which a pacemaker/implantable cardioverter-defibrillator (ICD) is indicated but not placed. Note: Patients who do have a pacemaker/ICD are allowed on study.
   8. Screening 12-lead ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) >500 msec. Note: Patients who have a pacemaker may be included regardless of calculated QTc interval.
   9. Supine systolic blood pressure <90 mm Hg, or symptomatic orthostatic hypotension, defined as a decrease in systolic blood pressure upon standing of >20 mmHg despite medical management (e.g., midodrine, fludrocortisones) in the absence of volume depletion.
8. Planned stem cell transplant. Note: Stem cell collection is permitted. Timing should be discussed with sponsor-investigator.
9. History of malignancy (other than AL amyloidosis) within 3 years before the date of study enrollment. Note: Exceptions are squamous and basal cell carcinomas of the skin, carcinoma in situ of the cervix or breast, or other non-invasive lesion that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 3 years).
10. For patients with known or suspected COPD, chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal are excluded. Note: FEV1 testing is required only for patients known or suspected of having COPD and patients must be excluded if FEV1 is < 50% of predicted normal.
11. Moderate or severe persistent asthma within the past 2 years, or currently has uncontrolled asthma of any classification. Note: Patients who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate.
12. Participant meets one of the following criteria:

    1. Known history of human immunodeficiency virus (HIV).
    2. Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen (HBsAg)). Note: Patients with resolved infection (i.e., patients who are HBsAg negative with antibodies to total hepatitis B core antigen (anti-HBc) with or without the presence of hepatitis B surface antibody (anti-HBs)) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. However, patients with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of HBV vaccination, do not need to be testing for HBV DNA by PCR, and will not be excluded.
    3. Seropositive for hepatitis C (except in the setting of a sustained virologic response (SVR), defined as aviremia at least 12 weeks after completion of antiviral therapy).
13. Concurrent medical condition or disease (e.g., active systemic infection) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study.
14. Has not recovered from adverse events due to prior anti-cancer therapy to <= grade 1 or baseline (other than alopecia).
15. Systemic treatment with any of the following within 7 days prior to the first dose of study drug:

    * Steroid therapy for anti-neoplastic intent
    * Known moderate or strong cytochrome P450 3A (CYP3A) inhibitors
    * Known moderate or strong CYP3A inducers ** Note: Patients who are taking strong CYP3A4 inducers must discontinue their use at least 5 half-lives prior to the first dose of study treatment
16. Administration or consumption of any of the following within 3 days prior to the first dose of study drug:

    * Grapefruit or grapefruit products
    * Seville oranges (including marmalade containing Seville oranges)
    * Starfruit
17. Patient anticipates use of prohibited medications or foods during study participation.
18. Major surgery within 2 weeks before Cycle 1 Day 1, or will not have fully recovered from surgery, or has surgery planned during the time the subject is expected to participate in the study or within 2 weeks after the last dose of study treatment administration.

    * Note: Patients with planned surgical procedures to be conducted under local anesthesia may participate.
19. Known or suspected of not being able to comply with the study protocol or the patient has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the patient (e.g., compromise their well-being) or that could prevent, limit, or confound the protocol-specified assessments.
20. Woman who is pregnant or breastfeeding or planning to become pregnant while enrolled in this study or within 3 months following discontinuation of daratumumab or venetoclax.
21. Have received vaccination with live attenuated vaccines within 4 weeks of first study agent administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with reported dose limiting toxicities (Phase 1) | Up to 1 cycle (1 cycle is equal to 28 days)
  A dose limiting toxicity (DLT) will be defined as an adverse event that are considered by the investigator to be at least possibly related to the study drugs and are observed within the DLT assessment window (Cycle 1, Days 1 to 28) except those that are clearly and incontrovertibly due to extraneous causes.
Maximum tolerated dose (MTD) (Phase 1) | Up to 1 cycle (1 cycle is equal to 28 days)
  The MTD is the last dose cohort at which no more than one instance of dose limiting toxicities (DLT) is observed among 6 participants treated. If the MTD cannot be determined due to lack of DLTs during the DLT window, the maximum dose level of venetoclax administered during the study will be declared the Recommended Phase 2 dose (RP2D).
Recommended phase 2 dose (RP2D) (Phase1) | Up to 1 cycle (1 cycle is equal to 28 days)
  If the MTD cannot be determined due to lack of DLTs during the DLT window, the maximum dose level of venetoclax administered during the study will be declared the Recommended phase 2 dose (RP2D).
Proportion of participants who achieve a complete hematologic response (CHR) (Phase 2) | Up to 2 years
  CHR is defined per updated 2021 International Society of Amyloidosis (ISA) consensus criteria as an absence of amyloidogenic light chains (either free and/or as part of a complete immunoglobulin) defined by negative immunofixation electrophoresis of both serum and urine, and also either a free-light chain (FLC) ratio within the reference range or the uninvolved FLC concentration is greater than involved FLC concentration with or without an abnormal FLC ratio. Participants with positive serum immunofixation (S-IFE) and confirmed daratumumab immunofixation (IFE) interference, that meet all other clinical criteria for CHR, will be considered CHR. CHR requires confirmation by 1 repeat assessment. Proportion and 95% binomial exact confidence interval will be reported

SECONDARY OUTCOMES:
Percentage of participants with treatment-emergent adverse events attributable to study treatment | Up to 2 years
  Percentage of participants with reported treatment-emergent adverse events by type, severity, and attribution of probably, possible, or related to study drugs, according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be reported for both phases of the study.
Proportion of participants with complete hematologic response (CHR) (Phase 2) | Up to 2 years
  CHR is defined per updated 2021 International Society of Amyloidosis (ISA) consensus criteria as an absence of amyloidogenic light chains (either free and/or as part of a complete immunoglobulin) defined by negative immunofixation electrophoresis of both serum and urine, and also either a free-light chain (FLC) ratio within the reference range or the uninvolved FLC concentration is greater than involved FLC concentration with or without an abnormal FLC ratio. Participants with positive serum immunofixation (S-IFE) and confirmed daratumumab immunofixation (IFE) interference, that meet all other clinical criteria for CHR, will be considered CHR. CHR requires confirmation by 1 repeat assessment.
Overall hematologic response rate (ORR) (Phase 2) | Up to 2 years
  The proportion of participants enrolled in Phase 2 who experience a hematologic objective response defined as a partial response (PR), a very good partial response (VGPR), or a complete response (CR) per updated 2021 ISA consensus criteria.
Organ response rate (orRR) (Phase 2) | Up to 2 years
  Organ disease considered to be quantifiable for response includes cardiac disease, renal disease, and hepatic disease. Liver organ response must be monitored by the ISA Consensus Criteria. Renal organ response must be monitored by Palladini criteria. Cardiac response must be monitored by the Boston University criteria. The proportion of participants enrolled in Phase 2 who experience an organ response (Heart, kidney, and/or liver).
Median Major Organ Deterioration Progression-Free Survival (MOD-PFS) (Phase 2) | Up to 2 years
  MOD-PFS is defined as the time that elapses between initiation of trial therapy and the earlier of hematologic disease progression, cardiac deterioration that requires cardiac transplant, left ventricular assist device, or intra-aortic balloon pump, end-stage renal disease that requires hemodialysis or renal transplant, or death from any cause for participants enrolled in Phase 2. Median survival times will be reported in months along with 95% confidence intervals obtained using the Brookmeyer and Crowley (1982) method.
Time to complete response (TTCR) (Phase 2) | Up to 2 years
  TTCR is defined as the time that elapses between the initiation of trial therapy (C1D1) and the first time that complete hematological response (CHR) is recorded for participants enrolled in Phase 2.
Median Time To Next Treatment (TTNT) (Phase 2) | Up to 2 years
  For the RP2D combination, TTNT is defined as the time that elapses between the initiation of study treatment (C1D1) to the time the participant initiates subsequent anti-cancer therapy for participants enrolled in Phase 2. Median time will be reported in months along with 95% confidence intervals.
Median Duration of response (DOR) (Phase 2) | Up to 2 years
  DOR is defined as the time that elapses between the day of first documented hematological response to trial therapy (PR or better whichever is first recorded) to the date of first documented evidence of hematological disease progression participants enrolled in Phase 2. Median duration will be reported in months along with 95% confidence intervals.
Median Progression-Free Survival (PFS) (Phase 2) | Up to 2 years
  PFS is defined as the time that elapses between initiation of trial therapy and the earlier of the day of first documented disease progression (either hematologic or organ) or death from any cause for participants enrolled in Phase 2. Median survival times will be reported in months along with 95% confidence intervals obtained using the Brookmeyer and Crowley (1982) method.
Median Overall Survival (OS) (Phase 2) | Up to 2 years
  The overall survival is defined as the time that elapses between the initiation of trial therapy (C1D1) and the date of death from any cause for all participants enrolled in Phase 2. Median survival times will be reported in months along with 95% confidence intervals obtained using the Brookmeyer and Crowley (1982) method.
Overall number of participant deaths (Phase 2) | Up to 2 years
  The number of participants enrolled in Phase 2 whose death occurred while the participant was on study will be reported.
Number of treatment-related mortalities (Phase 2) | Up to 2 years
  The number of participants enrolled in Phase 2 whose death was at least possibly attributable to treatment will be reported.
Proportion of participants with infection (Phase 2) | Up to 2 years
  The proportion of participants enrolled in Phase 2 who develop a documented infection will be reported.
Percentage of participants with a cardiac event (Phase 2) | Up to 2 years
  The percentage of participants enrolled in Phase 2 with a documented cardiac event will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Chung, MD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No